CLINICAL TRIAL: NCT03136003
Title: DDAVP vs Exercise in Patients With Mild Hemophilia A - Which is Better and do They Work Synergistically in Improving Hemostasis?
Brief Title: DDAVP vs. Exercise in Patients With Mild Hemophilia A
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Canadian Hemophilia Society (Other); Unity Health Toronto (Other); Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Manuel Carcao, Hematologist, The Hospital for Sick Children
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1000054948
Record Dates: First submitted 2017-04-27; First posted 2017-05-02 (Actual); Last update posted 2017-12-04 (Actual); Status verified 2017-11

CONDITIONS: Mild Haemophilia A Without Inhibitor
MeSH Terms: interventions — Deamino Arginine Vasopressin; Exercise

STUDY DESIGN:
Masking Description: The randomization of the participant to a study arm will be done prior to the study visit by the pharmacy at the hospital. The Investigator and study team will know the arm each participant is in before the patient's visit. This information will also be provided to the participant before the visit.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm A: DDAVP followed by exercise (Experimental): Intervention #1: DDAVP. The participant will take either 1 or 2 nasal sprays of IN DDAVP. For patients weighing <50 kg: 150 ug (i.e. 1 spray into one nostril) and patients weighing ≥50 kg: 300 ug (i.e. 2 sprays - one into each nostril).
  Intervention #2: Exercise
  Interventions: Drug: DDAVP; Behavioral: Exercise
- Arm B: DDAVP alone (Active Comparator): Intervention #1: DDAVP. The participant will take either 1 or 2 nasal sprays of IN DDAVP. For patients weighing <50 kg: 150 ug (i.e. 1 spray into one nostril) and patients weighing ≥50 kg: 300 ug (i.e. 2 sprays - one into each nostril).
  Intervention #2: no further intervention (rest)
  Interventions: Drug: DDAVP
- Arm C: Exercise alone (Experimental): Intervention #1: Exercise
  Intervention #2: no further intervention (rest)
  Interventions: Behavioral: Exercise
- ARM D: Exercise followed by DDAVP (Experimental): Intervention #1: Exercise
  Intervention #2: DDAVP. The participant will take either 1 or 2 nasal sprays of IN DDAVP. For patients weighing <50 kg: 150 ug (i.e. 1 spray into one nostril) and patients weighing ≥50 kg: 300 ug (i.e. 2 sprays - one into each nostril).
  Interventions: Drug: DDAVP; Behavioral: Exercise

INTERVENTIONS:
Drug: DDAVP — The participant will take either 1 or 2 nasal sprays of IN DDAVP (known as Octostim® in Canada). After receiving IN DDAVP, the participant will rest for 30 minutes.
  Other Names: IN DDAVP, Octostim
  Arms: ARM D: Exercise followed by DDAVP; Arm A: DDAVP followed by exercise; Arm B: DDAVP alone
Behavioral: Exercise — The participant will exercise on a stationary cycle-ergometer using the previously-validated, progressively-incremental Godfrey protocol. Per the Godfrey protocol, the participant starts cycling on the calibrated cycle-ergometer with an initial exercise load dependent on their height. The workload is increased every minute in standard increments also based on the participant's height. All participants will exercise until they complete 3-minutes of cycling at 85% of their maximum predicted heart rate or exhaustion (whichever is first). Upon completion of planned exercise, work load is decreased to zero watts and participants will continue cycling at this cool-down rate for an additional 3-minutes, before getting off the ergometer.
  Arms: ARM D: Exercise followed by DDAVP; Arm A: DDAVP followed by exercise; Arm C: Exercise alone

SUMMARY:
Individuals with mild hemophilia A (MHA) bleed infrequently but can in the setting of trauma which often is when participating in sports/exercise. Although both exercise and DDAVP (desmopressin) can raise Factor 8/Von Willebrand Factor (FVIII/VWF levels), it is not clear whether the pathophysiological mechanism is the same. Consequently it is not known if DDAVP and exercise would have additive effects in raising FVIII:C and VWF levels or if one would one negate the effect of the other. The aim of this 2 center (Sickkids and Columbus, Ohio), prospective, cross-over design study is to compare the impact of exercise vs. DDAVP on hemostasis in patients with MHA and also to investigate the impact of sequentially administering these interventions on their hemostatic indices.

DETAILED DESCRIPTION:
Persons with mild hemophilia A (MHA) (defined as having a FVIII level of >5% to ≈40%) bleed infrequently but can in the setting of trauma which can often is in the context of participating in sports/exercise. FVIII levels temporarily rise with stress, exercise and with DDAVP (1-desamino-8-D-arginine vasopressin, desmopressin). In the case of DDAVP, the Hospital for Sick Children (SickKids) Hemophilia Team and others have shown that FVIII and VWF levels rise by 2-4 fold with DDAVP. Consequently many persons with MHA in an attempt to reduce their risk of bleeding take intranasal (IN) DDAVP prior to sports activities/exercise. IN DDAVP is reasonably expensive ($300/bottle of Octostim® in Canada and $700/bottle of Stimate® in USA), requires fluid restriction, and may be associated with nausea, vomiting, seizures and tachyphylaxis.

Recently, our group completed a pilot/feasibility study to evaluate the impact of a prescribed, moderate intensity aerobic exercise regimen on hemostatic indices in 30 children with hemophilia A [HA] or B [HB] (all severities) and documented a significant improvement in multiple coagulation parameters (platelet count, FVIII:C and von Willebrand factor [VWF]) with exercise. This improvement was particularly pronounced in 13 post-adolescent males with mild-moderate HA. In this sub-cohort, we noted a mean 2.3 fold increase in FVIII:C immediately after exercise, which remained significantly elevated at 1.9 fold,1 hour after completion of exercise

These changes in hemostatic variables associated with aerobic exercise may be protective against bleeding, and may negate the need to administer IN DDAVP immediately prior to sports participation.

Although both exercise and DDAVP can raise FVIII/VWF levels, it is not clear whether the pathophysiological mechanism in which they do this is the same. Consequently it is not known if DDAVP and exercise would augment each other's effects in raising FVIII:C and VWF levels or if one would one negate the effect of the other. Herein, we propose a prospective, interventional study of exercise vs IN DDAVP in 40-50 post adolescent (13-21 yr) males with MHA to compare their impact on hemostasis and also to investigate the impact of sequentially administering these interventions on hemostatic indices.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥13 years of age and ≤21 years of age with Mild Hemophilia A (MHA), with a historical baseline FVIII:C level of ≥5% to ≤40% followed at either the Hospital for Sick Children or St. Michael's Hospital (Toronto).
* Patients ≥13 years of age and ≤21 years of age with genetically confirmed Mild Hemophilia A (MHA), with FVIII:C level of ≥5% to ≤50% followed at either the Hospital for Sick Children or St. Michael's Hospital (Toronto).

Exclusion Criteria:

* A currently circulating or history of a previous inhibitor ( ≥0.5 BU) within the past 5 years. As inhibitor development in MHA is rare, it is not expected that any patient will be excluded for this reason.
* Any FVIII infusion or DDAVP use in the preceding week. This is to avoid an residual FVIII still being present in a patient who has taken an extended half-life FVIII.
* Co-existence of a congenital bleeding disorder other than MHA (e.g. VWD).
* Prior history of coronary artery disease or pulmonary disease, severe arthropathy interfering with ability to exercise.
* Patients on beta-blockers, anti-platelet agents or regular non-steroidal anti-inflammatory medications (e.g. Celebrex).
* Patients with an active infectious or inflammatory condition. This includes HIV, active hepatitis B or C as reflected in elevated AST, ALT, RNA positivity for hepatitis B or C.
* Patients who are active (defined as smoking daily) smokers (cigarettes, marijuana). This exclusion is put into place as we do not know if daily smoking will impact on the hemostatic response to either exercise or DDAVP.
* Patients with limited exercise tolerance for any reason.
* Patients with a history of a recent bleed (in preceding 2 weeks) in any location, or a joint/muscle bleed in the lower limbs in the preceding 4 weeks.
* Patients who for medical reasons should not receive DDAVP [those with renal or CNS disease (e.g. brain tumor)] or have previously experienced adverse events with DDAVP (e.g. hypotensive event; seizure).

Ages: 13 Years to 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-07-04 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Factor 8 level after exercise | Baseline, 30 min post intervention #1, 30 min post intervention#2 and 90 minute post intervention#2
  To compare the increase in Factor 8 levels (FVIII:C) (measured as absolute and fold increase) associated with moderate intensity aerobic exercise (approximately 15 minutes of gradually increasing aerobic exercise culminating in 3-minutes of exercise at 85% of the predicted maximum heart rate) vs. IN DDAVP in post-adolescent males with MHA.

SECONDARY OUTCOMES:
Factor 8 level after sequential administration of exercise followed by IN DDAVP (or vice versa) | Baseline, 30 min post intervention #1, 30 min post intervention#2 and 90 minute post intervention#2
  To determine the absolute and fold increase in Factor 8 levels (FVIII:C) associated with the sequential administration of exercise followed by IN DDAVP (or vice versa).
Associations between baseline physical activity scores and Factor 8 levels after exercise | Baseline, 30 min post intervention #1, 30 min post intervention#2 and 90 minute post intervention#2
  To explore the impact of baseline physical activity (measured using the International Physical Activity Questionnaire [IPAQ]-short form) on exercise induced increase in Factor 8 levels (FVIII:C).

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Carcao, Principal Investigator — Staff Haematologist
Locations (2):
- Canada (2):
  - St. Michael's Hospital, Toronto, Ontario
  - The Hospital for Sick Children, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
To ensure the safety of patients and to confirm the validity of our hypothesis, we plan to:
  * Meet after the first 10 patients have completed the study.
  * Analyze data from first 10 patients. This includes safety data as well as results of the blood tests including the standard hemostasis testing (FVIII;C, VWF:Ag, VWF:RCo, VWF:CBA, VWF:pp), and platelet function (PFA).
  * Determine whether there are measurable outcomes justifying further enrollment and DSMB will be able to make recommendations regarding terminating the study or amending the protocol if they deem that there are safety issues.
  * If any of the first 10 subjects develops any unexpected medical complication we will suspend recruitment pending re-evaluation of the study by the DSMB.